CLINICAL TRIAL: NCT02668874
Title: A Clinical Trial Comparing Isolite® vs Cotton Roll Isolation in the Placement of Dental Sealants
Brief Title: A Clinical Trial Comparing Isolite® vs. Cotton Roll Isolation in the Placement of Dental Sealants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Iowa (Other)
Collaborators: Delta Dental of Iowa (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 201502801
Record Dates: First submitted 2015-11-10; First posted 2016-01-29 (Estimated); Results first posted 2022-02-01 (Actual); Last update posted 2022-02-01 (Actual); Status verified 2022-01

CONDITIONS: Dental Caries on Pit and Fissure Surface
Keywords: Pit and Fissure sealants; Isolation; permanent teeth; children; Isolite®; Dental caries
MeSH Terms: conditions — Van der Woude syndrome; Dental Caries

STUDY DESIGN:
Intervention Model Description: Simple randomization will be used for assignment of the treatment groups. Randomization: Two application methods will be used in each subject in order to place sealants, one using the Isolite system and one using the cotton roll system.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Triple:
  Participants, Investigator, and Outcome assessors do not know the randomization. However, it was hard to blind the care provider.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Isolite System (Other): The Isolite technique utilizes a flexible plastic dental adapter to separate the cheek and tongue prior to sealant placement.
  Interventions: Device: Isolite System
- Cotton Roll technique (Other): A cotton roll is placed between the cheek and tongue prior to sealant placement.
  Interventions: Other: Cotton Roll Technique

INTERVENTIONS:
Device: Isolite System
  Arms: Isolite System
Other: Cotton Roll Technique
  Arms: Cotton Roll technique

SUMMARY:
The purpose of this split-mouth, randomized, controlled trial is to evaluate the retention rates of sealants placed under Isolite vs. cotton roll isolation. This study will also compare the patient and operator acceptability and satisfaction of the two isolation techniques as well as the time consumed for sealant application during the two isolation techniques.

DETAILED DESCRIPTION:
104 regular patients at the College of Dentistry Department of Pediatric Dentistry Clinics, ages 6-16 years, will be invited to participate in this study. Matched contralateral pairs of first and second molars and premolars will be randomized to receive sealants with the use of the device (Isolite) for isolation or with the use of cotton roll isolation. All sealants will be placed by pediatric dentistry residents. Sealants will be placed on first and second permanent molars that have a matched contralateral molar requiring a sealant as well. Photographs may be taken of the sealants on the day of placement and at a 6-month and 12 month recalls. Retention of the sealants will be evaluated and scored by calibrated pediatric dentists.

ELIGIBILITY:
Inclusion Criteria:

* Healthy patients: American Society of Anesthesiologists (ASA) I or II
* Good cooperation: Frank1 3 or 4
* Aged between 6-16 years old at the day of sealant placement
* Minimum of two, maximum of sixteen, matched contralateral permanent molars or premolars.

Exclusion Criteria:

* Teeth with a history of past or current caries
* Teeth with a linical presentation of fluorosis, hypoplasia or any developmental anomalies
* Teeth with clinical or radiographic evidence of pathology
* Teeth with a history of restoration or sealant
* Patients who are poorly behaved

Ages: 6 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 104 (Actual)
Dates: Start 2015-02; Primary Completion 2017-08-21 (Actual); Study Completion 2017-08-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shin, Study Director — Director of Clinical Research
Locations (1):
- University of Iowa College of Dentistry and Dental Clinics, Iowa City, Iowa, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from the Pediatric Dentistry Clinic at the University of Iowa College of Dentistry and Dental Clinics.
Pre-assignment Details: Of the 104 enrolled subjects, 104 met the inclusion criteria and were randomized to treatment.
Units Other Than Participants: teeth
Groups:
- Cotton Roll System: A cotton roll is placed between the cheek and tongue prior to sealant placement.
Period: Overall Study
Arm/Group | Isolite System | Cotton Roll System
Started | 104; 203 teeth | 104; 203 teeth
6 Months After Placement | 59; 113 teeth | 59; 113 teeth
Completed | 47; 82 teeth | 47; 82 teeth
Not Completed | 57; 121 teeth | 57; 121 teeth

BASELINE CHARACTERISTICS:
Groups:
- Overall Group: The Isolite® technique differs in that it utilizes a flexible plastic dental adapter to separate the teeth from the cheek and tongue. The resident dentist will show the child the Isolite® before it is placed in the mouth. The resident with whom the child is scheduled will then apply the sealants.
  Isolite® technique: The Isolite technique utilizes a flexible plastic dental adapter to separate the cheek and tongue prior to sealant application.
Arm/Group | Overall Group
Number analyzed (Participants) | 103
Age, Continuous [Mean (Standard Deviation); unit: years] | 10.57 (3.12)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 48
  Male | 51
  Unknown | 4
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Sealant Retention Percentage at 12 Months After Treatment
Description: Physical examination will be done in order to determine if there is a percentage difference in retention rate of teeth, specifically 12 months after treatment.
Time Frame: 12 months after treatment
Measure: Count of Units; unit: teeth
Units Other Than Participants: teeth
Groups:
- Isolite® Technique Device: The Isolite® technique differs in that it utilizes a flexible plastic dental adapter to separate the teeth from the cheek and tongue. The resident dentist will show the child the Isolite® before it is placed in the mouth. The resident with whom the child is scheduled will then apply the sealants.
  Isolite® technique: The Isolite technique utilizes a flexible plastic dental adapter to separate the cheek and tongue prior to sealant application.
- Cotton Roll Technique Device: The resident dentist with whom the child is scheduled with apply the sealants after the cotton roll technique has been placed.
  Cotton Roll technique: A cotton roll is placed between the cheek and tongue prior to sealant application
Arm/Group | Isolite® Technique Device | Cotton Roll Technique Device
Number analyzed (Participants) | 47 | 47
Number analyzed (teeth) | 82 | 82
teeth | 59 | 66

ADVERSE EVENTS:
Time Frame: Adverse events were collected over a 12 month time-period
Description: no adverse events were reported
Arm/Group | Isolite® Technique Device | Cotton Roll Technique Device
All-Cause Mortality (participants affected / at risk) | 0/99 | 0/99
Serious Adverse Events (participants affected / at risk) | 0/99 | 0/99
Other Adverse Events (participants affected / at risk) | 0/99 | 0/99

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-09-01): https://cdn.clinicaltrials.gov/large-docs/74/NCT02668874/Prot_SAP_000.pdf